CLINICAL TRIAL: NCT04526691
Title: Phase 1b, Multicenter, Open-label Study of Datopotamab Deruxtecan (Dato-DXd) in Combination With Pembrolizumab With or Without Platinum Chemotherapy in Subjects With Advanced or Metastatic Non-Small Cell Lung Cancer (TROPION-Lung02)
Brief Title: Datopotamab Deruxtecan (Dato-DXd) in Combination With Pembrolizumab With or Without Platinum Chemotherapy in Subjects With Advanced or Metastatic Non-Small Cell Lung Cancer (TROPION-Lung02)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DS1062-A-U102; 2020-006047-25 (EudraCT Number); jRCT2031200193 (Other: JAPIC); KEYNOTE-B43 (Other: Merck Sharpe & Dohme LLC); MK-3475-B43 (Other: Merck Sharpe & Dohme LLC)
Record Dates: First submitted 2020-08-21; First posted 2020-08-26 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Advanced or Metastatic NSCLC
Keywords: Advanced or Metastatic NSCLC; Datopotamab deruxtecan (Dato-DXd); Pembrolizumab; KEYNOTE; DS-1062a
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Carboplatin; Cisplatin

STUDY DESIGN:
Intervention Model Description: Dose escalation and dose expansion model
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Datopotamab deruxtecan (Dato-DXd) (Experimental): Dose Escalation and Dose Expansion: Datopotamab deruxtecan (Dato-DXd) in combination with pembrolizumab with or without platinum chemotherapy in participants with advanced or metastatic NSCLC
  Interventions: Drug: Datopotamab deruxtecan; Drug: KEYTRUDA®; Drug: Carboplatin; Drug: Cisplatin

INTERVENTIONS:
Drug: Datopotamab deruxtecan — Intravenous infusion every 3 weeks (Q3W) on Day 1 of each 21-day cycle (starting datopotamab deruxtecan dose of 4.0 mg/kg)
  Other Names: Dato-DXd
Drug: KEYTRUDA® — Intravenous infusion Q3W on Day 1 of each 21-day cycle (fixed pembrolizumab dose 200 mg Q3W)
  Other Names: pembrolizumab
Drug: Carboplatin — Intravenous infusion Q3W on Day 1 or Day 2 of each 21-day cycle (AUC 5)
Drug: Cisplatin — Intravenous infusion Q3W on Day 1 or Day 2 of each 21-day cycle (75 mg/m^2)

SUMMARY:
This study will assess safety and treatment activity of datopotamab deruxtecan (Dato-DXd) in combination with pembrolizumab with or without platinum chemotherapy in participants with advanced or metastatic non-small cell lung cancer.

DETAILED DESCRIPTION:
The primary objective of this study will assess safety and treatment activity of datopotamab deruxtecan (Dato-DXd) in combination with pembrolizumab with or without 4 cycles of platinum chemotherapy in participants with advanced or metastatic NSCLC who have either been previously treated or are treatment naïve in a metastatic setting.

Two dose levels of Dato-DXd (4.0 mg/kg and 6.0 mg/kg) will be studied in combination with 200 mg fixed-dose pembrolizumab in 6 study cohorts. This study will be conducted sequentially and dose escalation will occur according to lower dose to higher dose in the same combination regimen (4.0 mg/kg to 6.0 mg/kg) and from 2-drug combination (Dato-DXd and pembrolizumab) to 3-drug combination regimen (Dato-DXd, pembrolizumab, and carboplatin or cisplatin).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed at diagnosis of NSCLC that:

  * Is advanced or metastatic.
  * Participants with non-squamous histology must have documented negative test results for actionable EGFR and ALK genomic alterations. Participants with squamous histology are required to undergo testing for EGFR and ALK genomic alterations if they are nonsmokers or under the age of 40 years.
  * Has either documented negative or unknown test results for actionable genomic alterations in ROS1, NTRK, BRAF, RET, MET, or other actionable oncogenic driver kinases.
  * Participants with tumors that harbor KRAS mutations are eligible for this study.
  * Participants with non-actionable genomic alterations in EGFR, ALK, ROS1, NTRK, BRAF, RET, MET, or other kinases are eligible for the study.
* Documentation of radiological disease progression while on or after receiving the most recent treatment regimen, if any, for advanced or metastatic NSCLC.
* Must meet the following prior therapy requirements for advanced or metastatic NSCLC:

  * Dose escalation (all cohorts): Has received ≤2 lines of prior anticancer therapy for locally advanced or metastatic NSCLC.
  * Dose expansion (cohorts with 4.0 mg/kg or 6.0 mg/kg Dato-DXd in combination with 200 mg fixed dose of pembrolizumab): Has not received PD-1/PD-L1, PD-L2, CTLA-4 directed immunotherapy and may or may not have been treated with systemic chemotherapy for advanced or metastatic NSCLC.
  * Dose expansion (cohorts with 4.0 mg/kg or 6.0 mg/kg Dato-DXd in combination with 200 mg fixed dose of pembrolizumab and 4 cycles of AUC 5 carboplatin or cisplatin 75 mg/m^2): Has not been treated with systemic anticancer therapy for advanced or metastatic NSCLC.
* Willing and able to undergo a mandatory tumor biopsy.
* Archival tumor tissue from initial diagnosis, to the extent that archival tumor tissue is available, for measurement of TROP2 expression levels or other biomarkers.
* Has adequate bone marrow reserve and organ function at baseline within 7 days prior to Cycle 1 Day 1.
* Is not a candidate for surgical resection or chemoradiation with curative intent.

Exclusion Criteria:

* Experienced grade 3 or higher immune-related adverse events (AEs) with prior treatment of anti-programmed cell death 1 (anti-PD-1), anti-programmed cell death ligand 1 (anti-PD-L1), or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
* Received a live vaccine within 30 days prior to the first dose of study treatment.
* Active, known, or suspected autoimmune disease.
* Concomitant use of chronic systemic (IV or oral) corticosteroids or other immunosuppressive medications, except for managing AEs.
* Prior organ transplantation, including allogeneic tissue or solid organ transplantation.
* Has spinal cord compression or clinically active central nervous system metastases, defined as untreated and symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms.
* History of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
* Clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses.
* History of another primary malignancy (beyond NSCLC) except for:

  * Malignancy treated with curative intent and with no known active disease for ≥3 years.
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
  * Adequately treated carcinoma in situ without evidence of disease.
  * Participants with a history of prostate cancer (tumor/node/metastasis stage) of Stage ≤T2cN0M0 without biochemical recurrence or progression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose-limiting Toxicities (DLTs) and Treatment-emergent Adverse Events (TEAEs) | Baseline up to Cycle 1 (Days 1 to 21) for DLTs and up to 28 days after last dose for TEAEs, up to approximately 30 months post-dose

SECONDARY OUTCOMES:
Objective Response Rate | Baseline up to BOR (confirmed CR or PR), up to approximately 30 months post-dose
Duration of Response | From first objective response (confirmed CR or PR) to PD or death (whichever occurs first), up to approximately 30 months post-dose
Progression-free Survival | Baseline up PD or death (whichever occurs first), up to approximately 30 months post-dose
Overall Survival | Baseline up to death (any cause), up to approximately 30 months post-dose
Pharmacokinetic Parameter Maximum Plasma Concentration (Cmax) of Dato-DXd, Total Anti-TROP2 Antibody, and MAAA-1181a | Cycle 1, Day 1: pre-dose, 30 minutes, 3 hours, 5 hours, and 7 hours post-dose; Cycles 1 and 3, Day 2, Day 4, Day 8, and Day 15; Cycles 2-4, Cycle 6, and Cycle 8, Day 1: pre-dose and post-dose (each cycle is 21 days)
Pharmacokinetic Parameter Time to Maximum Plasma Concentration (Tmax) of Dato-DXd, Total Anti-TROP2 Antibody, and MAAA-1181a | Cycle 1, Day 1: pre-dose, 30 minutes, 3 hours, 5 hours, and 7 hours post-dose; Cycles 1 and 3, Day 2, Day 4, Day 8, and Day 15; Cycles 2-4, Cycle 6, and Cycle 8, Day 1: pre-dose and post-dose (each cycle is 21 days)
Pharmacokinetic Parameter Area Under the Plasma Concentration-Time Curve (AUC) of Dato-DXd, Total Anti-TROP2 Antibody, and MAAA-1181a | Cycle 1, Day 1: pre-dose, 30 minutes, 3 hours, 5 hours, and 7 hours post-dose; Cycles 1 and 3, Day 2, Day 4, Day 8, and Day 15; Cycles 2-4, Cycle 6, and Cycle 8, Day 1: pre-dose and post-dose (each cycle is 21 days)
  Area under the plasma concentration-time curve up to last quantifiable time (AUClast) and area under the plasma concentration-time curve during dosing interval (AUCtau) will be assessed.
Anti-drug Antibodies for Dato-DXd and Pembrolizumab | Baseline up to approximately 30 months post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (24):
- United States (9):
  - Mayo Clinic, Scottsdale, Arizona
  - City of Hope, Duarte, California
  - Johns Hopkins Kimmel Cancer Center, Washington D.C., District of Columbia
  - Mayo Clinic, Jacksonville, Florida
  - Johns Hopkins Kimmel Cancer Center at Bayview, Baltimore, Maryland
  - The Skip Viragh Outpatient Cancer Building, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Quantum Santa Fe, Santa Fe, New Mexico
  - NEXT Oncology, San Antonio, Texas
- Italy (3):
  - Instituto Europeo Di Oncologica, Milan
  - Azienda Ospedaliera San Gerardo, Monza
  - Istituto Nazionale Tumori Fondazione G. Pascale di Napoli Struttura di Oncologia, Naples
- Japan (3):
  - National Cancer Center Hospital East, Chiba
  - National Cancer Center Hospital, Tokyo
  - Showa Medical University Hospital, Tokyo
- Spain (5):
  - H. Vall Hebrón (Vall Hebron Institut de Oncologia - VHIO), Barcelona
  - START Madrid - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - (CIOCC-START) Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Puerta de Hierro, Majadahonda
- Taiwan (4):
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital NCKUH, Tainan
  - National Taiwan University Hospital NTUH, Taipei

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/